CLINICAL TRIAL: NCT07291349
Title: Examination of the Effect of a Psychoeducational-Developmental Support Program on Adolescents' Relative Deprivation, Distress Levels, Peer Relationships, and Basic Psychological Needs
Brief Title: Effect of a Psychoeducational-Developmental Support Program on Adolescents' Relative Deprivation, Distress Levels, Peer Relations and Basic Psychological Needs
Acronym: PDSP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aziz Küçükkelepçe (Other)
Responsible Party: Sponsor-Investigator, Aziz Küçükkelepçe, Doctoral Researcher / PhD Candidate, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HÜ-EK-2024/13; HÜ-EK-2024/13 (Other: Hacettepe University)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Psychological Well-being
Keywords: Relative Deprivation; Distress-Eustress; Peer Relationships; Basic Psychological Needs; Psychoeducational-Developmental Intervention; Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive the Psychoeducational-Developmental Support Program delivered once per week for 11 weeks.
  Interventions: Behavioral: Psychoeducational-Developmental Support Program
- Control Group (No Intervention): Participants will receive no intervention during the study period. Pre-test and post-test assessments will be conducted.

INTERVENTIONS:
Behavioral: Psychoeducational-Developmental Support Program — The Psychoeducational-Developmental Support Program is an 11-week structured behavioral intervention developed through needs analysis with teachers. The program includes weekly sessions containing psychoeducational and developmental support activities designed to reduce distress-eustress imbalance, decrease relative deprivation, and strengthen peer relationships and basic psychological needs.
  Arms: Intervention Group

SUMMARY:
This study aims to examine the effectiveness of a Psychoeducational-Developmental Support Program on adolescents' distress-eustress levels, relative deprivation, peer relationships, and basic psychological needs. The program will be implemented with high school students using a pre-test/post-test control group design. The 11-week intervention includes structured psychoeducational and developmental activities. Assessments of distress-eustress, relative deprivation, peer relations, and basic psychological needs will be conducted before and after the intervention. A follow-up test will be administered one month later. The program is expected to produce significant improvements in adolescents' psychological and social functioning.

DETAILED DESCRIPTION:
This study investigates the effectiveness of an 11-week Psychoeducational-Developmental Support Program in reducing adolescents' distress-eustress levels and relative deprivation, while supporting peer relationship quality and the satisfaction of basic psychological needs. The program was developed based on a needs analysis conducted with teachers and incorporates structured psychoeducational content and developmental support activities tailored to adolescents.

The study employs a pre-test/post-test control group experimental design with high school students from three districts in Istanbul. The intervention group will receive weekly psychoeducational-developmental sessions, whereas the control group will receive no intervention. Measurements will include the Distress-Eustress Scale for Adolescents (Turkish Form), the Relative Deprivation Scale-Adolescent Form, the Peer Relations Scale, and the Basic Psychological Needs at School Scale. A retention assessment will be conducted one month after the intervention to evaluate the sustainability of the program's effects.

Data will be analyzed using the Mann-Whitney U test, the Wilcoxon Signed-Rank test, and effect size calculations (p < .05). The program is expected to lead to meaningful and lasting improvements in adolescents' emotional and psychosocial well-being.

ELIGIBILITY:
Inclusion Criteria: *High school students enrolled in selected schools in Istanbul.

* Aged 14-18 years.
* Able to participate in weekly psychoeducational-developmental sessions.
* Provide informed assent (and parental consent where required).

Exclusion Criteria: * Students with severe cognitive or developmental impairments that prevent participation.

* Students currently receiving psychological treatment specifically targeting distress or related constructs.
* Failure to obtain parental consent.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Distress-Eustress Levels | Baseline (pre-test) and post-intervention (11 weeks).
  Change in adolescents' distress-eustress levels from pre-test to post-test as measured by the Distress-Eustress Scale for Adolescents (Turkish Form). Higher distress scores indicate greater emotional strain; higher eustress scores indicate positive stress response.

SECONDARY OUTCOMES:
Relative Deprivation | Baseline and post-intervention (11 weeks).
  Change in adolescents' perceived relative deprivation measured by the Relative Deprivation Scale-Adolescent Form from pre-test to post-test. Higher scores indicate greater perceived deprivation.
Peer Relationships | Baseline and post-intervention (11 weeks).
  Change in adolescents' peer relationship quality measured by the Peer Relations Scale from pre-test to post-test. Higher scores indicate better peer relationship functioning.
Basic Psychological Needs at School | Baseline and post-intervention (11 weeks).
  Change in adolescents' satisfaction of basic psychological needs measured by the Basic Psychological Needs at School Scale from pre-test to post-test. Higher scores indicate greater need satisfaction.

OTHER OUTCOMES:
Retention of Program Effects | 1 month post-intervention
  One-month follow-up assessment administered to the experimental group to evaluate the persistence of intervention effects on distress-eustress, relative deprivation, peer relationships, and basic psychological needs.

CONTACTS AND LOCATIONS:
Overall Officials: Haktan Demircioğlu, Assoc. Prof. Dr., Study Director — Hacettepe University, Faculty of Health Sciences
Locations (1):
- Participating High Schools in Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared due to confidentiality requirements and restrictions specified by the ethics committee for underage participants.